CLINICAL TRIAL: NCT02931227
Title: Accuracy of Zero Heat Flux Cutaneous Temperature in Intensive Care Adults
Acronym: TempCore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TempCore
Record Dates: First submitted 2016-09-05; First posted 2016-10-13 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2016-09

CONDITIONS: Continuous Non Invasive Cutaneous Temperature; Zero Heat Flux Method; Esophageal Temperature; Arterial Temperature; Intracerebral Temperature

ARMS (4):
- Brain-injured group (Experimental)
  Interventions: Procedure: temperature obtained by the non-invasive method of zero-heat flux; Procedure: esophageal temperature; Procedure: intracerebral temperature
- Hypothermia group (Experimental)
  Interventions: Procedure: temperature obtained by the non-invasive method of zero-heat flux; Procedure: esophageal temperature; Procedure: intracerebral temperature
- Hyperthermia group (Experimental)
  Interventions: Procedure: temperature obtained by the non-invasive method of zero-heat flux; Procedure: esophageal temperature; Procedure: intracerebral temperature
- PICCO group (Experimental)
  Interventions: Procedure: temperature obtained by the non-invasive method of zero-heat flux; Procedure: esophageal temperature; Procedure: intracerebral temperature; Procedure: arterial temperature

INTERVENTIONS:
Procedure: temperature obtained by the non-invasive method of zero-heat flux
Procedure: esophageal temperature
Procedure: intracerebral temperature
Procedure: arterial temperature
  Arms: PICCO group

SUMMARY:
Temperature is one of the vital signs usually monitored in patients of ICUs. Indeed, fever occurs frequently in ICU especially in brain injured patients and may require targeted temperature management (TTM) in special case as intracranial hypertension or post cardiac arrest. In ICU, non invasive device to monitor temperature are not recommended and only invasive ones are accurate enough for TTM. Arterial pulmonary temperature is still the gold standard, but esophageal device is currently used in ICU patients.

The goal of this study is to compare accuracy of a continuous noninvasive cutaneous temperature using zero-heat-flux (ZHF) method to esophageal temperature, arterial temperature and intracerebral temperature if present for clinical monitoring.

All adults patients admitted in the neurosurgical or surgical ICU are eligible for inclusion into this study.

Assessment of temperature will be continuously monitored by esophageal probe (MON-A-THERM, 12Fr, COVIDIEN, Dublin, Ireland) (Teso), ZHF sensor (SpotOn, 3M, St Paul, MN, USA) (TZHF) and, in patients requiring cardiac output monitoring, by femoral arterial catheter (Pulsiocath PICCO, PULSION, Munich, Germany) (Tart). The correct positioning of the esophageal probe will be controlled by chest X-ray. The ZHF temperature sensor (TZHF) will be placed on the forehead as recommend by the manufacturer and connected to the SpotOn monitor. Intra cerebral temperature (Tbrain) will be obtained with an intracranial probe used as calibrator for partial pressure of O2 in brain (PbO2, Licox®Combined Oxygen and Temperature Probe 462 mm device necessary for monitoring severe brain injured patients. The ZHF sensor will be changed every 24 hours according to the manufacturer's directions for use. Temperatures will be recorded automatically at a 5-minutes interval via the patient's monitor with an electronic data acquisition system (Data Collect, Phillips) for a maximum of 5 days.

For each patient included, data recorded will be: demographic and clinical particulars for each patient; information on hemodynamics, sedative, analgesic and inotropic agents, use of neuromuscular blockades and their indication, reason of hypo or hyperthermia (spontaneous or therapeutic), indication and the means used (neuromuscular blockades, external or internal cooling) in case of Targeted Temperature Management; complications related to the ZHF sensor application.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old
* patients who required core temperature monitoring

Exclusion Criteria:

* front disrepair
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Comparison a continuous non-invasive cutaneous temperature using zero-heat flux method | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France